CLINICAL TRIAL: NCT02862171
Title: A Follow-On, Open-Label Trial To Assess Continued Safety Of And Adherence To The Dapivirine (25 Mg) Vaginal Ring-004 In Healthy, HIV-Negative Women
Brief Title: To Assess Continued Safety of and Adherence to the Dapivirine (25 mg) Vaginal Ring-004 in Healthy, HIV-negative Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IPM 032
Record Dates: First submitted 2016-07-25; First posted 2016-08-10 (Estimated); Results first posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: HIV Prevention
MeSH Terms: interventions — Dapivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dapivirine Vaginal Ring-004 (Experimental): Dapivirine Vaginal Ring, 25 mg.Each participant will engage in the screening process for up to 45 days prior to enrolment and will use the monthly Dapivirine Vaginal Ring for a period of up to 12 months. IPM will have the option to extend this trial period.
  Interventions: Drug: Dapivirine Vaginal Ring-004

INTERVENTIONS:
Drug: Dapivirine Vaginal Ring-004 — To assess the safety profile of the 25 mg Dapivirine Vaginal Ring-004, when inserted at monthly intervals, in an open-label trial
  Other Names: TMC-120

SUMMARY:
A follow-on, open label trial to assess continued safety of and adherence to the Dapivirine(25mg) vaginal ring-004 in healthy, HIV-negative women

DETAILED DESCRIPTION:
Phase IIIb, multicenter follow-on open-label trial to evaluate the continued adherence to and safety of the DVR, inserted at monthly intervals by healthy, HIV negative women who had participated in the IPM 027 Phase III DVR trial. All women who participated in IPM 027 (NCT 01539226) and were HIV-negative at screening for IPM 032, were eligible.

Participants who provided written informed consent at screening were invited to undergo screening assessments for the trial. The Enrollment Visit had to occur within 45 days after the Screening Visit. Note: In the event that participation in IPM 027 was stopped prematurely and IPM 032 was activated at the RC, the IPM 027 Last Product Use Visit (LPUV) and the IPM 032 Screening and Enrollment Visits could be combined for participants who were eligible to enroll in IPM 032.

All participants received the DVR containing 25 mg dapivirine at the Enrollment Visit, and attended a visit at the RC, 1 month after enrollment. Following this visit, a participant could continue on a 3 monthly visit schedule, at the Investigator's discretion. Monthly visits could, however, be extended up to the first 3 months of participation. From then on, all participants needed to switch to a 3-monthly schedule. Once the 3-monthly trial visit schedule commenced, three rings were dispensed at each visit. One ring was self-inserted at the RC and two additional rings were dispensed for the participant to take home, or dispensing took place as arranged with the participant.

The protocol made provision for at least 12 months of DVR use (with the LPUV scheduled at Month 12), which could also have been extended. Participants could continue with ring use past Month 12 and the RCs could continue scheduling the 3-monthly visits as per the participant visit schedule. Exit Visits of participants who completed 12 months or more on the trial commenced in October 2017 and ended in January 2019. Participants who were still enrolled in the trial in October 2017 and those who had been enrolled at a later stage in the trial were scheduled to attend the Month 12 Visit, irrespective of their visit schedule assignments. Exit Visits were then scheduled as per protocol, ie, 1 to 2 months after the Month 12 Visit. Exit Visits were optional for participants who discontinued early from the trial.

Adherence assessments included analysis of dapivirine residual levels in returned used rings, correlation analysis of dapivirine residual levels with visual inspection of used rings, and self-reported acceptability and adherence.

The HIV-1 incidence and the occurrence of HIV-1 drug resistance were assessed using HIV rapid testing and genotyping, respectively.

Social and behavioral parameters were assessed qualitatively and quantitatively. Quantitative assessments included evaluation of the feasibility of 3-monthly follow-up visits and evaluation of the proportion of participants undergoing unscheduled HIV rapid tests (ie, in between the scheduled 3 monthly follow-up visits).

Safety assessments included adverse event (AE) reporting, safety laboratory assessments, pregnancy testing, physical examination, vital sign assessments, pelvic examination, sexually transmitted infection (STI) tests, cervical cytology, and assessments of social harms.

Throughout the trial, all participants received pre- and post-test HIV counseling, HIV/STI risk reduction counseling, and contraceptive, condom and vaginal ring adherence counseling.

ELIGIBILITY:
Inclusion Criteria:

Women must meet all the following criteria to be eligible to enrol in the trial:

1. Previously enrolled in the IPM 027 trial
2. Available for all visits and consent to follow all procedures scheduled for the trial
3. Using an effective method of contraception at the Enrolment Visit, and intending to use an effective contraceptive method for the duration of trial participation, unless post-menopausal with no history of menses for one year prior to screening
4. HIV-negative as determined by the HIV algorithm applied at Screening/Pre- Enrolment
5. Willing to refrain from participation in another research trial using drugs, vaccines, medical devices and microbicides for the duration of the IPM 032 trial
6. Willing to provide adequate locator information for trial retention purposes and be reachable per local standard procedures (e.g., by home visit or telephone; or via family or close neighbour contacts); confidentiality to be maintained.

Exclusion Criteria:

Women who meet any of the following criteria are NOT eligible to enrol in the trial:

1. Investigational product use permanently discontinued in response to an AE (where the AE was considered related to investigational product) or safety-related concern while taking part in the IPM 027 trial
2. Participant self-report of taking post-exposure prophylaxis (PEP) within ≤ 2 months at Screening Visit Note: Participants may be enrolled after completing the PEP regimen and a negative HIV test was documented at least 2 months prior to screening for IPM 032
3. Currently pregnant, intends to become pregnant or currently breast-feeding
4. Known drug abuse or alcohol dependence in the 12 months prior to screening
5. Participated in another research trial (other than IPM 027) using drugs, medical devices, microbicides or oral pre-exposure prophylaxis agents within 30 days prior to screening
6. Any new illness or condition(s), chronic condition(s) or abnormal laboratory finding(s) that, in the opinion of the investigator, might put the participant at risk, or interfere with the trial objectives or the participant's adherence to trial requirements

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 941 (Actual)
Dates: Start 2016-07-12 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Steytler, Study Director — International Partnership for Microbicides
Locations (6):
- South Africa (5):
  - Qhakaza Mbokodo, Ladysmith, KwaZulu-Natal
  - MatCH Research Unit, Pietermaritzburg, KwaZulu-Natal
  - Madibeng Centre for Research, Brits, North West
  - Desmond Tutu HIV Foundation, Cape Town, Western Cape
  - Ndlovu Medical Centre, Elandsdoorn
- MRC/UVRI Uganda Research Unit on AIDS, Entebbe, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Steytler J, Craig C, van der Ryst E, Van Baelen B, Nuttall J, van Niekerk N, Mellors J, Parikh U, Wallis C; Ring Study and the DREAM Trial Study Teams. Characterization of Viruses in Phase 3 and Phase 3b Trials (the Ring Study and the Dapivirine Ring Extended Access and Monitoring Trial) of the Dapivirine Vaginal Ring for Human Immunodeficiency Virus Type 1 Infection Risk Reduction. Clin Infect Dis. 2023 Mar 21;76(6):996-1002. doi: 10.1093/cid/ciac875. PMID 36345569
- [Derived] Nel A, van Niekerk N, Van Baelen B, Malherbe M, Mans W, Carter A, Steytler J, van der Ryst E, Craig C, Louw C, Gwetu T, Mabude Z, Kotze P, Moraba R, Tempelman H, Gill K, Kusemererwa S, Bekker LG, Devlin B, Rosenberg Z; DREAM Study Team. Safety, adherence, and HIV-1 seroconversion among women using the dapivirine vaginal ring (DREAM): an open-label, extension study. Lancet HIV. 2021 Feb;8(2):e77-e86. doi: 10.1016/S2352-3018(20)30300-3. PMID 33539761

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Up to 1,400 former IPM 027 participants were to be enrolled at 6 Research Centres (RC) - 5 RCs in SA and one RC in Uganda.
Pre-assignment Details: Overall, 1,034 participants who had participated in IPM 027 were screened for inclusion in IPM 032 open-label trial. Of these, 941 (941/1,034; 91.0%) participants were enrolled, and 848 (848/941; 90.1%) participants completed the trial. Of the 941 enrolled participants, 150 rolled over directly from IPM 027, without any interruption in DVR use.
Groups:
- Dapivirine Vaginal Ring-004: Dapivirine Vaginal Ring, 25 mg.Each participant will engage in the screening process for up to 45 days prior to enrolment and will use the monthly Dapivirine Vaginal Ring for a period of up to at least 12 months.
  Dapivirine Vaginal Ring-004: To assess the safety profile of the 25 mg Dapivirine Vaginal Ring-004, when inserted at monthly intervals, in an open-label trial
Period: Overall Study
Arm/Group | Dapivirine Vaginal Ring-004
Started | 941
Completed | 848
Not Completed | 93
Not completed — Death | 1
Not completed — Lost to Follow-up | 13
Not completed — Withdrawal by Subject | 57
Not completed — Non-compliance | 4
Not completed — HIV-1 seroconversion | 18

BASELINE CHARACTERISTICS:
Population: Healthy, HIV-negative women who had participated in IPM 027
Arm/Group | Dapivirine Vaginal Ring-004
Number analyzed (Participants) | 941
Age, Customized [Mean (Standard Deviation); unit: years]
  18 - 45 years | 30.1 (6.32)
Sex: Female, Male [Count of Participants; unit: Participants] — DVR, inserted at monthly intervals by healthy, HIV-negative women who had participated in the IPM 027 Phase III DVR trial. All women who participated in IPM 027 and were HIV-negative at screening for IPM 032, were eligible.
  Participants
    Female | 941
    Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Sub-Saharan Africa is most strongly affected by the HIV/AIDS epidemic; 53% (approximately 19.6 million people) of the global total living with HIV in 2017 were in this region.
  Sub-Saharan Africa accounted for 44% (approximately 800,000 people) of the global total of new HIV infections and 40% (approximately 380,000 people) of the global total of deaths from HIV/AIDS-related illnesses in 2017.
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 931
    White | 0
    More than one race | 10
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Women from South Africa and Uganda were enrolled.
  participants
    South Africa | 820
    Uganda | 121

OUTCOME MEASURES:

1. Primary Outcome: The Safety Profile of the 25 mg Dapivirine Vaginal Ring-004, When Inserted at Monthly Intervals. Participants Attended RC at Monthly Visits (up to Max of Three Monthly Visits) Followed by 3-monthly Follow-up Visits.
Description: Safety assessments included adverse event (AE) reporting; all product-related AEs, Grade 3 or 4 AEs, SAEs.
Time Frame: at least 12 months and up to 17 months
Population: The safety population included all participants who were enrolled, and received and inserted at least one DVR.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapivirine Vaginal Ring-004
Number analyzed (Participants) | 941
Participants
  At least one treatment emergent adverse event (TEAE) | 616
  At least one serious TEAE | 20
  At least one serious non-TEAE | 3
  At least one DAIDS Grade 3 or 4 TEAE | 37
  At least one product-related TEAE | 6
  TEAEs leading to death | 1
  TEAEs leading to temporary IP discontinuation | 2
  Urogenital TEAEs | 410
  Social harms reported as TEAEs | 8
  Non-TEAEs | 31

2. Primary Outcome: Adherence to the Use of the 25 mg Dapivirine Vaginal Ring-004 Inserted at Monthly Intervals, in an Open-label Trial
Description: Determined dapivirine residual amounts in returned used vaginal rings.
Time Frame: at least 12 months and up to 17 months
Population: The safety population included all participants who were enrolled, and received and inserted at least one DVR.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Dapivirine Vaginal Ring-004
Number analyzed (Participants) | 941
mg
  Enrollment. The month the ring was used is defined as the month the ring was dispensed. | 20.77 (1.271)
  Trial Month 1. The month the ring was used is defined as the month the ring was dispensed. | 20.57 (1.453)
  Trial Month 2.The month the ring was used is defined as the month the ring was dispensed. | 20.59 (1.478)
  Trial Month 3. The month the ring was used is defined as the month the ring was dispensed. | 20.83 (1.513)
  Trial Month 4. The month the ring was used is defined as the month the ring was dispensed | 20.61 (1.503)
  Trial Month 5. The month the ring was used is defined as the month the ring was dispensed | 20.70 (1.448)
  Trial Month 6. The month the ring was used is defined as the month the ring was dispensed. | 20.77 (1.406)
  Trial Month 7. The month the ring was used is defined as the month the ring was dispensed | 20.44 (1.445)
  Trial Month 8. The month the ring was used is defined as the month the ring was dispensed. | 20.59 (1.446)
  Trial Month 9.The month the ring was used is defined as the month the ring was dispensed. | 20.72 (1.583)
  Trial Month 10. The month the ring was used is defined as the month the ring was dispensed. | 20.47 (1.575)
  Trial Month 11. The month the ring was used is defined as the month the ring was dispensed. | 20.82 (1.626)
  Trial Month 12. The month the ring was used is defined as the month the ring was dispensed | 20.84 (1.459)
  Trial Month 13. The month the ring was used is defined as the month the ring was dispensed | 20.49 (1.371)
  Trial Month 14. The month the ring was used is defined as the month the ring was dispensed. | 20.81 (1.355)
  Trial Month 15. The month the ring was used is defined as the month the ring was dispensed. | 20.92 (1.668)
  Trial Month 16. The month the ring was used is defined as the month the ring was dispensed. | 20.20 (1.273)

3. Secondary Outcome: Incidence of HIV-1 Seroconversion
Description: Rapid and specialised laboratory testing according to a pre-specified HIV testing algorithm
Time Frame: at least 12 months and up to 17 months
Population: This population excluded all participants who were included in the safety population but who were found to have been HIV-1 infected at the Enrollment Visit (ie, participants who had seroconverted after enrollment but were retrospectively found to be HIV-1 infected at enrollment).
Measure: Number; unit: events per 100 person-years
Arm/Group | Dapivirine Vaginal Ring-004
Number analyzed (Participants) | 938
events per 100 person-years | 1.8

4. Secondary Outcome: Number of Participants Who Acquired HIV-1 With HIV-1 Drug Resistance-associated Mutations. Infection
Description: Viral genotype (including NGS) resistance testing methods which include sensitive methods to detect low frequency drug-resistant variants.
Time Frame: at least 12 months and up to 17 months
Population: The virology population included all HIV infected participants in the m-ITT population, with the exception of those participants who seroconverted after LPUV. That is, participants who were HIV-1 RNA negative at LPUV, and who became infected after LPUV, were excluded. Genotypic analyses from the small numbers of participants with infection at enrollment, or with no detectable HIV-1 RNA at the LPUV but with seroconversion at the Exit Visit, were described individually.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapivirine Vaginal Ring-004
Number analyzed (Participants) | 18
Participants | 5

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a minimum period of 12 months and a maximum of 17 months per participant. Treatment-emergent adverse events were defined as AEs which occurred/worsened after the first insertion of the IP, up to 6 weeks after last ring use.
Arm/Group | Dapivirine Vaginal Ring-004
All-Cause Mortality (participants affected / at risk) | 1/941
Serious Adverse Events (participants affected / at risk) | 20/941
Other Adverse Events (participants affected / at risk) | 616/941
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapivirine Vaginal Ring-004 (N=941)
Stab wound, ankle fracture, fibula fracture, muscle strain, soft tissue injury, thermal burn (Injury, poisoning and procedural complications) | 7 (7)
Meningitis tuberculous, Pyelonephritis, Sepsis, vuval abscess (Infections and infestations) | 4 (4)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Hypertension, Hypertensive crisis (Vascular disorders) | 2 (2)
Sudden death (General disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapivirine Vaginal Ring-004 (N=941)
Infections (Infections and infestations) | 462 (462) — Upper respiratory tract infection, genital infection female, vulvovaginitis, genitourinary tract gonococcal infection, trichomoniasis, bacterial vaginosis, vulvovaginal candidiasis, viral rhinitis
Reproductive system (Reproductive system and breast disorders) | 197 (197) — Cervical dysplasia, vulvovaginal pruritus, dysmenorrhoea, pelvic pain
Headache (Nervous system disorders) | 33 (51)
Gastritis (Gastrointestinal disorders) | 28 (105)
Back pain (Musculoskeletal and connective tissue disorders) | 26 (73)
Hypertension (Vascular disorders) | 19 (20)

LIMITATIONS AND CAVEATS:
Interpretation of the HIV-1 incidence rates is limited by the lack of a concurrent placebo group in IPM 032.

Dapivirine residual levels in returned used rings do not provide adherence information at the time of potential exposure to and infection with HIV, eg, if a participant temporarily removes the DVR during sexual intercourse.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol: Protocol 2.0 Amendment 4.0 (2019-10-17): https://cdn.clinicaltrials.gov/large-docs/71/NCT02862171/Prot_000.pdf
  • Study Protocol: Protocol 2.0 Amendment 2.0 (2017-01-16): https://cdn.clinicaltrials.gov/large-docs/71/NCT02862171/Prot_001.pdf
  • Study Protocol: Protocol 2.0 Amendment 1.0 (2015-10-22): https://cdn.clinicaltrials.gov/large-docs/71/NCT02862171/Prot_002.pdf
  • Statistical Analysis Plan (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/71/NCT02862171/SAP_003.pdf